CLINICAL TRIAL: NCT04743908
Title: Community Network-driven COVID-19 Testing and Vaccination of Vulnerable Populations in the Central US (C3)
Brief Title: Community Network-driven COVID-19 Testing and Vaccination of Vulnerable Populations in the Central US
Acronym: C3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Howard Brown Health Center (Other); Community Action Place, Inc. (Other); Indiana University (Other); University of Arkansas (Other); Better Community Development, Inc. (Industry); Capitol Area Reentry Program Inc. (Industry); University of Texas Southwestern Medical Center (Other); San Jose State University (Other); George Mason University (Other); NORC at the University of Chicago (Other); Northwestern University (Other); Project Vida (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB20-1494; 3UG1DA050066-02S1 (NIH)
Record Dates: First submitted 2021-02-05; First posted 2021-02-08 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: Criminal Justice Involved; Latinx; Social Network Strategy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Using a two-arm randomized controlled trial design, participants will be enrolled into the SNS arm (involves social networking referrals only) or the SNS+messaging arm. The latter includes affirmation/misinformation correction messaging (discussion tools and coaching).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Network Strategy (SNS Condition) (No Intervention): Study staff will describe the Social Network Strategy, construct a plan for successfully referring network members into the study, and discuss compensation for the recruitment efforts. Study staff will specifically discuss network members of interest: "friend, family, coworker or someone you spend time with on a regular basis". Walkthrough and scenario play will be strategies to assist with planning regarding: (1) how the conversation will be raised, (2) how potential barriers to testing will be addressed, (3) how the screening by phone or web survey will be conducted, (4) how network members will have the option to bring others into the study visit with them, (5) what information about the study will be shared.
- Social Network Strategy + Messaging (Experimental): Study staff will describe the Social Network Strategy, construct a plan for successfully referring network members into the study, and discuss compensation for the recruitment efforts. Study staff will specifically discuss network members of interest: "friend, family, coworker or someone you spend time with on a regular basis". Walk through and scenario play will be strategies to assist with planning regarding: (1) how the conversation will be raised, (2) how potential barriers to testing will be addressed, (3) how the screening by phone or web survey will be conducted, (4) how network members will have the option to bring others into the study visit with them, (5) what information about the study will be shared. Finally, community developed COVID-19 public health messages will be shared in the participant's preferred language.
  Interventions: Other: Social Network Strategy + COVID-19 messaging

INTERVENTIONS:
Other: Social Network Strategy + COVID-19 messaging — Contextually adapted and theory-driven messages - misinformation correction and self-affirmation - to increase awareness, self-efficacy and community engagement in our adapted Social Network testing Strategy (SNS). SNS is an evidence-based testing intervention that has been widely used in multiple settings with marginalized individuals (ie substance-users) who facilitate the recruitment of their social contacts into testing services.
  Arms: Social Network Strategy + Messaging

SUMMARY:
This C3 project, Community network-driven COVID-19 testing of vulnerable populations in the Central US, will implement and evaluate a COVID-19 testing and vaccination approach that combines an evidence-based Social Network Testing Strategy (SNS) with community developed COVID-19 public health messages (SNS+). C3 will engage two disenfranchised populations across rural and urban sites in states across the Central US (Texas (TX), Louisiana (LA), Arkansas (AR), Indiana (IN), Illinois (IL)). C3 leverages NIDA's Justice Community Opioid Innovation Network (JCOIN), the PIs' extensive community located COVID-19 testing programs, and a network of established community partnerships. The collaborative community-academic partnerships, research and engagement infrastructure, and team's leadership across JCOIN will ensure that C3 can rapidly recruit, enroll and test most disenfranchised community members, (n=2400) and through this process, accelerate any forthcoming COVID-19 public health prevention interventions. C3 focuses on two communities most impacted by COVID-19: 1) Criminal justice involved (CJI) - non-incarcerated people with previous history of arrest/jail/prison, probation/parole, drug-court attendance, witnessed or experienced a negative interaction with police or law enforcement; and 2) Low-income Latinx - community members at 250% or below Federal Poverty Level. Both of these diverse populations, and the overlap between them, have some of the highest rates of COVID-19 infection and death in the United States. Messaging that affirms individual agency and corrects misinformation, combined with accessible and acceptable testing, is required to accelerate COVID-19 prevention for these populations.Using a two-arm randomized controlled trial design, participants will be enrolled into the Social Network testing Strategy (SNS) arm (involves social networking referrals only) or the Social Network testing Strategy with COVID-19 prevention messages (SNS+) messaging arm. The latter includes affirmation/misinformation correction messaging (discussion tools and coaching). SNS and SNS+messaging arms will both include an initial group of index study participants who will refer their network members into the study and the process will repeat itself one more time for a total of 3 waves. Indexes will refer network members (1st degree) and then those network members will refer one more round (2nd degree).

ELIGIBILITY:
Inclusion criteria:

Index community members will be:

1. 18 years or older (15-28 years old at University of Indiana site);
2. spend majority of their time in the metropolitan area or county where recruited;
3. have access to a phone for 21-day follow-up call; and
4. primary communication in English or Spanish (based on site; Spanish language for Howard Brown/Project Vida and UTSW) AND at least one of the following: (i) ever had CJI (operationalized as any jail, prison, arrest, parole (completed), probation, drug court); (ii) ever had negative interaction with police or law enforcement that did not lead to an arrest or jail/prison time (operationalized as ever stopped, searched, physically or verbally abused, or had another negative interaction with police or law enforcement); (iii) ever witnessed a negative interaction with police or law enforcement (iv) lower-income Latinx (operationalized as at or below 250% of FPL) (Not applicable for University of Indiana).

Social network referrals will be:

1. linked to the index as a "friend, family, coworker or someone you spend time with on a regular basis";
2. visit within two weeks of index visit;
3. 18 years or older;
4. spend the majority of their time in the metropolitan area or county where recruited;
5. have access to a phone for 21-day follow-up call; and
6. primary communication in English or Spanish.

Exclusion Criteria:

1. inability to provide informed consent; and
2. active COVID-19 symptoms per the Centers for Disease Control and Prevention (CDC). Participants with COVID-19 symptoms will be referred for free testing at existing partners for each of the study sites.
3. currently on parole
4. for the University of Indiana site, currently in foster care, on house arrest, on probation, detained at a federal facility or had a police encounter during which the officer(s) either asked for some form of identification and/or issued a traffic ticket, but did not have other CJI involvement.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1328 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Schneider, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Social Network Strategy (SNS Condition) | Social Network Strategy + Messaging
Started | 661 | 667
Completed | 478 | 485
Not Completed | 183 | 182
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 181 | 180
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Network Strategy (SNS Condition) | Social Network Strategy + Messaging | Total
Number analyzed (Participants) | 661 | 667 | 1328
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (14.8) | 39.7 (14.4) | 39.6 (14.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Assigned Sex at Birth: Female | 353 | 328 | 681
  Assigned Sex at Birth: Male | 296 | 329 | 625
  Assigned Sex at Birth: Intersex | 3 | 1 | 4
  Assigned Sex at Birth: Unknown, Refused, or Missing | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 213 | 217 | 430
  Not Hispanic or Latino | 427 | 429 | 856
  Unknown or Not Reported | 21 | 21 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 8 | 19
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 256 | 273 | 529
  White | 220 | 237 | 457
  More than one race | 31 | 24 | 55
  Unknown or Not Reported | 130 | 114 | 244
Self-Reported COVID-19 Tests at Baseline [Count of Participants; unit: Participants]
  Yes, participant had been tested for COVID-19 prior to baseline. | 530 | 519 | 1049
  No, participant had not been tested for COVID-19 prior to baseline. | 118 | 135 | 253
  Don't know, participant did not know if they been tested for COVID-19 prior to baseline. | 6 | 11 | 17
  Missing | 7 | 2 | 9
Self-Reported COVID-19 Vaccination at Baseline [Count of Participants; unit: Participants]
  Yes, participant reported that they have been vaccinated for COVID-19 | 479 | 471 | 950
  No, participant reported that they have not been vaccinated for COVID-19 | 173 | 182 | 355
  Don't know, participant didn't know whether they had been vaccinated for COVID-19 | 5 | 10 | 15
  Missing | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Tests Among Network Members Referred for COVID Testing (Network Tested).
Description: Network tested is measured at the participant level by the number of network members that are tested through the SNS.
Time Frame: 21 days from initial study visit for each participant
Measure: Count of Participants; unit: Participants
Arm/Group | Social Network Strategy (SNS Condition) | Social Network Strategy + Messaging
Number analyzed (Participants) | 661 | 667
Participants
  Tested | 444 | 437
  Not Tested | 196 | 206
  Missing Testing Data | 21 | 24

2. Primary Outcome: Total Number of Vaccinations Among Study Participants Given COVID Vaccine Information (Number Vaccinated)
Description: Number vaccinated is measured at the participant level by the number of study participants that are vaccinated through the SNS.
Time Frame: 21 days from initial study visit for each participant
Measure: Count of Participants; unit: Participants
Arm/Group | Social Network Strategy (SNS Condition) | Social Network Strategy + Messaging
Number analyzed (Participants) | 182 | 196
Participants
  Vaccinated | 18 | 27
  Not Vaccinated | 81 | 94
  Missing, Unknown, or Refused | 83 | 75

ADVERSE EVENTS:
Time Frame: 21 days from initial study visit for each participant
Arm/Group | Social Network Strategy (SNS Condition) | Social Network Strategy + Messaging
All-Cause Mortality (participants affected / at risk) | 1/661 | 2/667
Serious Adverse Events (participants affected / at risk) | 1/661 | 0/667
Other Adverse Events (participants affected / at risk) | 0/661 | 0/667
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Social Network Strategy (SNS Condition) (N=661) | Social Network Strategy + Messaging (N=667)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT04743908/Prot_SAP_000.pdf